CLINICAL TRIAL: NCT07032038
Title: First In Human, Multi-Center Open-Label Randomized Trial to Assess Safety of Rincell-1 Otic Neural Progenitor Cell-Based Therapy and Standard Care vs Standard Care Alone, in Adults With Neural Hearing Loss Eligible for Cochlear Implantation
Brief Title: First In Human Randomised Trial of Rincell-1 in Adults With a Cochlear Implant
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rinri Therapeutics (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1-25
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Sensorineural Hearing Loss; Presbyacusis; Auditory Neuropathy
Keywords: neural hearing loss; presbycusis; ANSD; auditory neuropathy; cell therapy; first in human
MeSH Terms: conditions — Hearing Loss, Sensorineural; Presbycusis; Auditory neuropathy; Retrocochlear Diseases | interventions — Cochlear Implantation

STUDY DESIGN:
Masking Description: Trial statistician, primary and secondary outcomes assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Unilateral CI + Rincell-1 (Experimental): Routine unilateral cochlear implantation with simultaneous single dose of Rincell-1
  Interventions: Drug: Otic neural progenitors; Device: cochlear implantation
- Standard Care Unilateral CI only (Active Comparator): Routine unilateral cochlear implantation only
  Interventions: Device: cochlear implantation

INTERVENTIONS:
Drug: Otic neural progenitors — Advanced Cell Therapy - tissue engineered product
  Arms: Standard Care Unilateral CI + Rincell-1
Device: cochlear implantation — cochlear implant

SUMMARY:
Rinri Therapeutics is conducting a clinical trial of a new cell therapy called Rincell-1. Rincell-1 is being developed to treat adults with neural hearing loss, either age related hearing loss or auditory neuropathy, who also meet criteria for a cochlear implant. The goals of this study are:

* To learn about the safety profile of Rincell-1, the procedure used to inject it and the medications given to promote the growth of the cells
* To evaluate how well Rincell-1 works by measuring changes in the function of auditory neurons.
* To understand if Rincell-1 can be easily and successfully given at the same time as cochlear implant surgery

Participants will be randomly assigned to one of two groups: one group that receives a standard care cochlear implant, and the other that will receive an injection of Rincell-1 at the same time as their standard care cochlear implant. Researchers will compare the safety of Rincell-1 in combination with a cochlear implant to a cochlear implant on its own.

Participants will take part in the trial for 52 weeks after CI surgery. During that time, they will have regular follow-ups and will take daily measurements at home of their hearing health.

DETAILED DESCRIPTION:
The proposed study is a Phase I/IIa, randomized, open-label, multi-center, First In Human trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) to investigate the safety of Rincell-1 as a treatment for neural hearing loss.

All participants will be recruited from adult patients who have been assessed as being eligible to receive a unilateral cochlear implant (CI) on the National Health Service at a UK CI Centre.

Trial participants will meet UK NICE criteria for cochlear implantation, and will be:

* Cohort 1: Patients with hearing loss due to bilateral progressive presbycusis (aged-related hearing loss)
* Cohort 2: Patients with postsynaptic Auditory Neuropathy Participants will be randomized (3:2), by cohort, to receive either Standard Care unilateral CI plus a single dose of Rincell-1 administered at the same time as CI surgery, or Standard Care unilateral CI alone. Each cohort will have up to a total of 10 participants: 6 in the CI+Rincell-1 arm, and 4 in the standard care CI arm. A total of up to 12 participants across the two cohorts will be dosed with Rincell-1.

Subjects will be followed up to 52 weeks post-implantation.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 Only

* Aged 60-74 years (inclusive) at time of screening
* Hearing Loss due to bilateral progressive presbycusis
* Approved for unilateral cochlear implantation as per UK NICE criteria (TA566)
* Documented threshold of ≥70dB in both ears at 1000, 2000 and 4000 Hz, and ≥50dB in both ears at 500 Hz, at time of eligibility

Cohort 2 Only

* Aged 18-74 years (inclusive) at time of screening
* Postsynaptic AN characterized by:

  * normal outer hair cell function evidenced by normal CM response, and aberrant or absent ABRs
  * disparity between relatively preserved pure-tone audiometric thresholds and significantly impaired speech perception abilities, in individuals who do not receive adequate benefit from acoustic HAs
  * genetic testing does not indicate a known synaptic dysfunction
* Approved for unilateral cochlear implantation as per UK NICE criteria TA566 and NHS England SSC1442

All participants (Cohort 1 and Cohort 2)

* Any gender
* Capable and willing to provide written informed consent
* History, examination and pre-operative imaging suggesting a healthy middle ear in the ear to be implanted, and a structurally normal and fully patent cochlea with no evidence of a widened vestibular aqueduct
* Both ears deemed suitable for cochlear implantation
* Pre-operative imaging suggesting adequate access for surgical approach for the injection of Rincell-1
* Willingness to be implanted with an Advanced Bionics HiRes Ultra 3D CI and suitable as per device IFU indication
* A MoCA-HI score of >24
* English speaker with sufficient comprehension and expressive language to complete questionnaires and speech tests

Exclusion Criteria:

Cohort 2 Only

• ECochG measurements and genetic testing suggestive of synaptopathy, including but not limited to: Otoferlin, CABP2, SLC17A8, KARS2, DIAPH3, GJB2, OPA1, or SLC52 A2 and A3 mutations.

All participants (Cohort 1 and Cohort 2)

* History of prelingual hearing loss
* History of hearing loss caused by infection or head trauma
* History of previous cochlear implantation, in either ear
* Documented hearing loss secondary to ototoxic medications
* Suspected or confirmed hearing loss that is wholly or partly unexplained by anatomic or physiologic abnormalities (non-organic hearing loss)
* Evidence of current conductive hearing loss defined as 20dB or greater average air-bone gap over three of the following frequencies: 500, 1000, 2000, 3000 or 4000 Hz
* History of diagnosed sudden SNHL, Ménière's disease, otosclerosis, cholesteatoma, acoustic neuroma, meningitis or confirmed/suspected autoimmune inner ear disease
* In the ear to be implanted, evidence of anatomical or morphological issues apparent on pre-operative imaging including inner, middle and outer ear malformations (including evidence of a hypoplastic/absent auditory nerve and/or bony/absent IAM) and any known factor that may restrict full insertion of the electrode array or injection of Rincell-1
* Any known contraindications or concerns about medical fitness for cochlear implantation surgery and the additional surgical steps required for Rincell-1 injection (including BMI ≥35) Any known contraindications or concerns about suitability for any of the trial medicinal products (refer to section 5.2, the IB, NIMP manual (Protocol Appendix 1) and relevant SmPCs)
* Diagnosis of active, moderate to severe autoimmune disorders or any immune disorder requiring immunosuppression in the past 5 years
* History of documented severe/significant allergic reaction that required treatment
* Malignancy under current active treatment or previous malignancy considered at substantial risk for progression or recurrence during trial interval, as determined by the Investigator
* Previous or current CNS neoplasms or head and neck cancer
* Previous recipient of a gene therapy, any other type of ATIMP, cell or organ transplantation, or recipient of multiple blood transfusions within the past 5 years
* Unable to be imaged using X-ray and/or MRI (including having any other implanted medical device that is MRI conditional)
* Currently pregnant or breastfeeding
* Unwilling to follow contraception requirements of the trial
* Current or future participation in another interventional research study or any hearing-related research study during the course of trial participation
* Diagnosis of any syndrome, disorder or disease that is auditory, neurological, neurocognitive, psychological or developmental in nature (including speech and language disorders and dyslexia) which, in the Investigator's judgement, could impact the trial assessments
* Any other reason, medical or otherwise, which, in the Investigator's judgment, could interfere with the participant's compliance with the protocol (including undertaking of daily objective testing) or interpretation of the study results, makes participating difficult or burdensome for the participant or compromises participant safety

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of AEs | From baseline (at screening) to 52 weeks post-implantation
  Frequency and severity of AEs considered related to Rincell-1 alone, the procedure used to administer Rincell-1, and to the CI device and/or the administered concomitant NIMP regime.

SECONDARY OUTCOMES:
Changes in mean ECAP thresholds | From post-implantation baseline to 40 weeks post-implantation
  Change from baseline to primary evaluation timepoint in mean ECAP threshold, measured at each electrode for each participant
Feasibility of administration of Rincell-1 | At time of administration
  Evaluated in terms of:
  * On-time delivery to theatre of the DP
  * Successful in-theatre DP preparation
  * Injection of the full DP into the target anatomical structure
  * DP sterility and viability

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hartley, Principal Investigator — Rinri Therapeutics
Locations (3):
- United Kingdom (3):
  - University Hospitals Birmingham, Birmingham
  - Cambridge University Hospital, Cambridge
  - Guy's and St Thomas' Trust, London

IPD SHARING:
Plan to Share IPD: No